CLINICAL TRIAL: NCT03037723
Title: Prospective Trial of Prone Whole-Breast RadiationTherapy Versus Supine Whole-Breast Radiation Therapy With and Without Respiratory Gating, a Dosimetric Comparison
Brief Title: Prone Whole-Breast RadiationTherapy Versus Supine Whole-Breast Radiation Therapy Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Anna Shapiro, Associate Professor, State University of New York - Upstate Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 496516
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer, Respiratory Gating, Prone
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prone/Supine Simulation (Other): It is institutional policy to perform CT simulation in left-sided breast cancer patients with and without the respiratory gating (this is one CT scan), in the face-up position. It is also standard of care to perform the face-down CT simulation in large breasted women. Both of these simulations are meant to reduce the exposure of the heart and lungs to radiation. In this study, all left-sided breast cancer patients that consent will receive face-up CT simulation with and without gating AND face-down CT simulation, regardless of breast size; thus, each patient is their own control.
  Interventions: Other: CT simulation

INTERVENTIONS:
Other: CT simulation

SUMMARY:
Radiation therapy to the breast has remained a standard practice for breast conserving therapy. Because of the location of the heart and lungs when patients are positioned face-up, whole breast radiation therapy has been reported to increase the risk of damage to the heart a few years after treatment until at least 20 years after exposure, and may affect cardiovascular mortality. Also, patients receiving whole breast radiation therapy are at an increased risk for development of secondary lung malignancies. Recent studies have demonstrated a significant reduction in dose to the heart and lungs when treated in the face-down position. Similarly, correcting for the movement of breathing (respiratory gating) in the face-up position has also become an available option for reducing unwanted dose to the heart and lungs, particularly in left sided breast cancers. No study to date has compared these newer organ-sparing techniques head-to-head for early stage breast cancer.

It is institutional policy to perform CT simulation in left-sided breast cancer patients with and without the respiratory gating (this is one CT scan), in the face-up position. It is also standard of care to perform the face-down CT simulation in large breasted women. Both of these simulations are meant to reduce the exposure of the heart and lungs to radiation.

In this study, all left-sided breast cancer patients that consent will receive face-up CT simulation with and without gating AND face-down CT simulation, regardless of breast size; thus, each patient is their own control.

The treating physician will determine which of the two simulations, if any, offers better protection to each patients' heart and lungs. Two dosimetrists will be required to independently verify planned dosimetry with all treatment setups. Treatment will be planned in standard fashion using the best of the two plans.

DETAILED DESCRIPTION:
Radiation therapy to the breast has remained a standard practice for breast conserving therapy. Because of the location of the heart and lungs when patients are positioned face-up, whole breast radiation therapy has been reported to increase the risk of damage to the heart a few years after treatment until at least 20 years after exposure, and may affect cardiovascular mortality. Also, patients receiving whole breast radiation therapy are at an increased risk for development of secondary lung malignancies. Recent studies have demonstrated a significant reduction in dose to the heart and lungs when treated in the face-down position. Similarly, correcting for the movement of breathing (respiratory gating) in the face-up position has also become an available option for reducing unwanted dose to the heart and lungs, particularly in left sided breast cancers. No study to date has compared these newer organ-sparing techniques head-to-head for early stage breast cancer.

It is institutional policy to perform CT simulation in left-sided breast cancer patients with and without the respiratory gating (this is one CT scan), in the face-up position. It is also standard of care to perform the face-down CT simulation in large breasted women. Both of these simulations are meant to reduce the exposure of the heart and lungs to radiation. In this study, all left-sided breast cancer patients that consent will receive face-up CT simulation with and without gating AND face-down CT simulation, regardless of breast size; thus, each patient is their own control.

The treating physician will determine which of the two simulations, if any, offers better protection to each patients' heart and lungs. Two dosimetrists will be required to independently verify planned dosimetry with all treatment setups. Treatment will be planned in standard fashion using the best of the two plans.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0-IIA left, breast cancer,
* After lumpectomy or segmental mastectomy,
* With negative surgical margins

Exclusion Criteria:

* Right breast cancer
* Positive surgical margins
* Stage 2B or higher

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-09; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
mean heart dose | immediate
  dosimetric parameter

CONTACTS AND LOCATIONS:
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darby SC, McGale P, Taylor CW, Peto R. Long-term mortality from heart disease and lung cancer after radiotherapy for early breast cancer: prospective cohort study of about 300,000 women in US SEER cancer registries. Lancet Oncol. 2005 Aug;6(8):557-65. doi: 10.1016/S1470-2045(05)70251-5. PMID 16054566
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Background] Deutsch M, Land SR, Begovic M, Wieand HS, Wolmark N, Fisher B. The incidence of lung carcinoma after surgery for breast carcinoma with and without postoperative radiotherapy. Results of National Surgical Adjuvant Breast and Bowel Project (NSABP) clinical trials B-04 and B-06. Cancer. 2003 Oct 1;98(7):1362-8. doi: 10.1002/cncr.11655. PMID 14508821
- [Background] Ng J, Shuryak I, Xu Y, Clifford Chao KS, Brenner DJ, Burri RJ. Predicting the risk of secondary lung malignancies associated with whole-breast radiation therapy. Int J Radiat Oncol Biol Phys. 2012 Jul 15;83(4):1101-6. doi: 10.1016/j.ijrobp.2011.09.052. Epub 2012 Jan 13. PMID 22245205
- [Background] Lymberis SC, deWyngaert JK, Parhar P, Chhabra AM, Fenton-Kerimian M, Chang J, Hochman T, Guth A, Roses D, Goldberg JD, Formenti SC. Prospective assessment of optimal individual position (prone versus supine) for breast radiotherapy: volumetric and dosimetric correlations in 100 patients. Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):902-9. doi: 10.1016/j.ijrobp.2012.01.040. Epub 2012 Apr 9. PMID 22494590
- [Background] Qi XS, Hu A, Wang K, Newman F, Crosby M, Hu B, White J, Li XA. Respiration induced heart motion and indications of gated delivery for left-sided breast irradiation. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):1605-11. doi: 10.1016/j.ijrobp.2011.01.042. Epub 2011 Apr 12. PMID 21489710